CLINICAL TRIAL: NCT02158351
Title: Role and Pathogenetic Mechanisms of Intestinal Microbiota in Non-alcoholic Fatty Liver Disease Severity in Obese and Non-obese Subjects
Brief Title: Gut Microbiota and Modulation of Liver Damage in NAFLD
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, STEFANO GINANNI CORRADINI, MD, PhD, University of Roma La Sapienza
Other Study IDs: 2943/14.11.2013
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Simple Steatosis (SS); Non-alcoholic Steatohepatitis (NASH); Obesity
Keywords: Simple steatosis (SS); Non-alcoholic steatohepatitis (NASH); Gut microbiota (GM); Non alcoholic fatty liver disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Liver Extracts

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool samples, serum, plasma, liver and (only in the obese patients) adipose tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Simple steatosis: We will run a cross-sectional observational study including two groups of human subjects: patients with simple steatosis (SS) or non-alcoholic steatohepatitis (NASH). Grouping in patients SS or NASH will be performed based on the histological diagnosis of the type of NAFLD obtained at operation (sleeve gastrectomy or cholecystectomy). BMI will be considered as a confounding variable to be statistically analyzed. Main hypothesis: GM can lead to liver inflammation in patients with liver fat accumulation.
  Interventions: Procedure: liver and white adipose tissue biopsies
- Non-alcoholic steato-hepatitis: We will run a cross-sectional observational study including two groups of human subjects: patients with simple steatosis (SS) or non-alcoholic steatohepatitis (NASH). Grouping in patients SS or NASH will be performed based on the histological diagnosis of the type of NAFLD obtained at operation (sleeve gastrectomy or cholecystectomy). BMI will be considered as a confounding variable to be statistically analyzed. Main hypothesis: GM can lead to liver inflammation in patients with liver fat accumulation.
  Interventions: Procedure: liver and white adipose tissue biopsies

INTERVENTIONS:
Procedure: liver and white adipose tissue biopsies

SUMMARY:
Several experimental data suggest that gut-derived endotoxin and GM composition can act as a "second hit" or insult to convert hepatic SS to NASH and cause both local hepatic and systemic inflammation.This study's aim is to analyze microbiota diversity, providing information both on intestinal microbial composition and on the metabolic processes linked to them. In addition, we will correlate, for the first time, GM composition to hepatic and white adipose tissue gene expression patterns of interest and serum and fecal markers possibly related to impaired fat storage and inflammation. We aim to provide preliminary data to design future intervention studies with pre- or probiotics or bile acid derivatives to prevent/treat inflammation and fibrosis in NAFLD patients.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) includes benign hepatic simple steatosis (SS) and the more severe steatohepatitis (NASH), which is characterized by inflammation and fibrosis potentially leading to cirrhosis and hepatocellular carcinoma. Current research is focused on what are the risk factors and determinants of NASH. NAFLD is associated with the metabolic syndrome, and the prevalence has been described to be up to 98% in morbidly obese individuals undergoing bariatric surgery. NAFLD in non-obese subjects have a different clinical profile than in obese individuals, being associated with insulin resistance (IR), differential distribution of visceral adipose tissue, recent increase in body weight and/or presence of overweight, intake of high cholesterol diet and genetic background.

Gut microbiota (GM) regulates fat metabolism in mice. In humans its alterations have been linked to diabetes, obesity, IR, atherosclerosis and inflammation, SS and NAFLD.

Several experimental data suggest that gut-derived endotoxin and GM composition can act as a "second hit" or insult to convert hepatic SS to NASH and cause both local hepatic and systemic inflammation. With regard to human studies, Muozaki et al. have recently showed, by using a polymerase chain reaction (PCR) TaqMan system approach, that obese patients with NASH, have a lower percentage of fecal Bacteroidetes (Bacteroidetes to total bacteria counts) compared to both SS and healthy controls and a higher percentage of C. coccoides compared to those with SS . In addition, Zhu et al. showed in pediatric subjects, by using a 16S ribosomal RNA detection method, an unique pattern of enterotypes in patients with NASH, in obese individuals with no sign of liver damage and in lean healthy controls. Finally, Wai-Sun Wong et al. showed, also using a 16S ribosomal RNA detection method, that a small group of Chinese NASH patients demonstrated fecal dysbiosis but not significant changes in biodiversity compared to healthy subjects. Finally, inflammation in patients with symptomatic atherosclerosis has been shown to be associated with lower levels of butyrate producing gut bacteria such as Roseburia.

Among the possible factors involved in determining NAFLD severity, serum bile acid (BA) concentration and its post-prandial variations have been recently linked to the regulation of body weight, liver fat and inflammation and glucose and lipid metabolism. These BA regulatory functions are mediated by their interaction with the farnesoid X receptor (FXR)and the G Protein-Coupled BA Receptor 1 (GPBAR1 or TGR5) at both hepatic and subcutaneous adipose tissue levels. No human study has been directed to investigating the mechanisms through which GM composition influences inflammation and fibrosis in both obese and non-obese patients with NAFLD.

Liver biopsy is clinically advisable during bariatric surgery, due to the high prevalence of NAFLD and NASH in morbidly obese patients. It has been previously suggested that the high prevalence of histologically proven NAFLD in patients with gallstones may also justify routine liver biopsy during cholecystectomy, even in non-obese subjects, to establish the diagnosis, stage, and possible therapy. The latter suggestion has been very recently reinforced by the evidence that, in humans, cholecystectomy may represent an independent risk factor for NAFLD detected at ultrasounds and by the experimental demonstration that cholecystectomy increases hepatic triglycerides content.

In the present research project we will study patients with histologically proven SS or with NASH. Liver biopsy will be performed during bariatric surgery (sleeve gastrectomy) or cholecystectomy in patients with preoperative evidence of NAFLD at ultrasounds. We will compare GM composition using, for the first time, the most accurate method available, that is metagenomic shotgun. This method allows to analyze microbiota diversity, providing information both on intestinal microbial composition and on the metabolic processes linked to them. In addition, we will correlate, for the first time, GM composition to hepatic and, only in the obese patients, also to white adipose tissue gene expression patterns of interest and serum and fecal markers possibly related to impaired fat storage and inflammation. We aim to provide preliminary data to design future intervention studies with pre- or probiotics or bile acid derivatives to prevent/treat inflammation and fibrosis in NAFLD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, equal or over 18 years old
2. Eligible for Sleeve Gastrectomy for obesity with BMI 35-50 kg/m2
3. Eligible for Cholecystectomy for symptomatic gallstones and bright liver at ultrasounds
4. Alcohol consumption is less than 20 g/d

Exclusion Criteria:

1. Having liver disease of other etiology
2. Having advanced liver disease
3. Having abnormal coagulation or other reason contraindicating a Liver Biopsy
4. On regular intake of medications known to cause or exacerbate steatohepatitis or antibiotic, pre- or probiotics in the previous 3 months
5. Use of vitamin E or fish oil supplements in the previous 2 months
6. Alcohol consumption of more than 20 g/dl
7. Inflammatory bowel diseases
8. previous gastrointestinal surgery modifying the anatomy (prior to bariatric surgery)
9. Pregnancy or lactating state

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: two groups of patients with morbid obesity undergoing sleeve gastrectomy will be enrolled. Grouping in patients with simple steatosis (SS) or non-alcoholic steatohepatitis (NASH) will be performed based on the histological diagnosis of the type of NAFLD obtained at operation. Two groups of non-obese patients undergoing cholecystectomy for gallstone disease will be enrolled. Grouping in patients with simple steatosis (SS) or non-alcoholic steatohepatitis (NASH) will be performed based on the histological diagnosis of the type of NAFLD obtained at operation.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
gut microbiota composition | 12 months
  In patients with simple steatosis SS vs those with NASH the gut microbiota composition is different even after BMI normalization

SECONDARY OUTCOMES:
In each patient group overall gut microbiota composition, and hepatic and (only in the obese patients submitted to bariatric surgery) adipose tissue mRNA expression of relevant lipid and inflammatory response pathways | 12 months
  In each patient group [simple steatosis (SS) and NASH], overall gut microbiota composition, and hepatic and (only in patients submitted to bariatric surgery) adipose tissue messenger ribonucleic acid (mRNA) expression of relevant lipid and inflammatory response pathways: Acetyl-coenzyme A-carboxylase (ACC1), Fatty acid Synthase (FAS), Sterol regulatory element-binding protein (SREBP1c), apolipoprotein B (ApoB), farnesoid X receptor (FXR), Carbohydrate-responsive element-binding protein (ChREBP), TGR5, Sterol regulatory element-binding protein (SREBP2a), liver X receptor (LXR), 3-hydroxy-3-methylglutaryl coenzyme A reductase (HMGCR), low density lipoprotein receptor (LDLR) , Proprotein-convertase-subtilisin/kexin type 9 (PCSK9), tumor necrosis factor α (TNF-α), toll-like receptor 4 (TLR-4), NLRP3 (NOD-like receptor 3), c-Jun N-terminal kinase (JUN-K)
In each patient group overall gut microbiota composition, and hepatic and (only in the obese patients submitted to bariatric surgery) adipose tissue mRNA expression of relevant lipid and inflammatory response pathways | 12 months
  In each patient group [simple steatosis (SS) and NASH], overall gut microbiota composition, and hepatic and (only in patients submitted to bariatric surgery) adipose tissue mRNA expression of relevant lipid and inflammatory response pathways: ACC1 (Acetyl-CoA carboxylase), FAS (Fatty acid Synthase), SREBP1c (Sterol regulatory element-binding protein), ApoB (apolipoprotein B), FXR (farnesoid X receptor), ChREBP (Carbohydrate-responsive element-binding protein), TGR5, SREBP2a (Sterol regulatory element-binding protein), LXR (liver X receptor), HMGCR (3-hydroxy-3-methylglutaryl coenzyme A reductase), LDLR (low density lipoprotein receptor) , PCSK9 (Proprotein Convertase Subtilisin/Kexin type 9), TNF-α (tumor necrosis factor α), TLR-4 toll-like receptor 4), NLRP3 (NOD-like receptor 3), JUN-K (c-Jun N-terminal kinase)

OTHER OUTCOMES:
In each group, overall gut microbiota composition, and serum fasting and (only in the obese patients) post-prandial bile acid levels, serum markers of inflammation and liver damage and white adipose tissue mRNA expression of relevant genes | 18 months
  In each patient group [simple steatosis (SS) and NASH], overall gut microbiota composition, and serum fasting and (only in patients submitted to bariatric surgery) post-prandial bile acid levels.In each patient group [simple steatosis (SS) and NASH], overall gut microbiota composition, and serum markers of inflammation and liver damage (endotoxin, TNF-alfa, IL-6, aspartate aminotransferase (AST), alanine aminotransferase (ALT), cytokeratin 18.In each patient group [simple steatosis (SS) and NASH], overall gut microbiota composition and white adipose tissue mRNA expression of relevant genes chosen on the base of the mRNA expression results on liver specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ginnani Corradini, MD, PhD, Study Director — Department of Translational and Precision Medicine, "Sapienza", University of Rome; Fredrik Backhed, PhD, Study Director — Wallenberg laboratoriet, Gotebörg, Sweden; Frida Leonetti, MD, PhD, Principal Investigator — University of Roma La Sapienza; Gianfranco Silecchia, MD, Principal Investigator — University of Roma La Sapienza; Francesco Gossetti, MD, Principal Investigator — University of Roma La Sapienza; Adriano De Santis, MD, Principal Investigator — University of Roma La Sapienza; Claudio Di Cristofano, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Stefano Ginanni Corradini, Rome, Italy

REFERENCES:
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Yilmaz Y. NAFLD in the absence of metabolic syndrome: different epidemiology, pathogenetic mechanisms, risk factors for disease progression? Semin Liver Dis. 2012 Feb;32(1):14-21. doi: 10.1055/s-0032-1306422. Epub 2012 Mar 13. PMID 22418884
- [Background] Backhed F, Manchester JK, Semenkovich CF, Gordon JI. Mechanisms underlying the resistance to diet-induced obesity in germ-free mice. Proc Natl Acad Sci U S A. 2007 Jan 16;104(3):979-84. doi: 10.1073/pnas.0605374104. Epub 2007 Jan 8. PMID 17210919
- [Background] Karlsson FH, Tremaroli V, Nookaew I, Bergstrom G, Behre CJ, Fagerberg B, Nielsen J, Backhed F. Gut metagenome in European women with normal, impaired and diabetic glucose control. Nature. 2013 Jun 6;498(7452):99-103. doi: 10.1038/nature12198. Epub 2013 May 29. PMID 23719380
- [Background] Ley RE, Turnbaugh PJ, Klein S, Gordon JI. Microbial ecology: human gut microbes associated with obesity. Nature. 2006 Dec 21;444(7122):1022-3. doi: 10.1038/4441022a. PMID 17183309
- [Background] Musso G, Gambino R, Cassader M. Gut microbiota as a regulator of energy homeostasis and ectopic fat deposition: mechanisms and implications for metabolic disorders. Curr Opin Lipidol. 2010 Feb;21(1):76-83. doi: 10.1097/MOL.0b013e3283347ebb. PMID 19915460
- [Background] Spencer MD, Hamp TJ, Reid RW, Fischer LM, Zeisel SH, Fodor AA. Association between composition of the human gastrointestinal microbiome and development of fatty liver with choline deficiency. Gastroenterology. 2011 Mar;140(3):976-86. doi: 10.1053/j.gastro.2010.11.049. Epub 2010 Dec 1. PMID 21129376
- [Background] Frazier TH, DiBaise JK, McClain CJ. Gut microbiota, intestinal permeability, obesity-induced inflammation, and liver injury. JPEN J Parenter Enteral Nutr. 2011 Sep;35(5 Suppl):14S-20S. doi: 10.1177/0148607111413772. Epub 2011 Aug 1. PMID 21807932
- [Background] Chassaing B, Etienne-Mesmin L, Gewirtz AT. Microbiota-liver axis in hepatic disease. Hepatology. 2014 Jan;59(1):328-39. doi: 10.1002/hep.26494. Epub 2013 Nov 15. PMID 23703735
- [Background] Mouzaki M, Comelli EM, Arendt BM, Bonengel J, Fung SK, Fischer SE, McGilvray ID, Allard JP. Intestinal microbiota in patients with nonalcoholic fatty liver disease. Hepatology. 2013 Jul;58(1):120-7. doi: 10.1002/hep.26319. Epub 2013 May 14. PMID 23401313
- [Background] Zhu L, Baker SS, Gill C, Liu W, Alkhouri R, Baker RD, Gill SR. Characterization of gut microbiomes in nonalcoholic steatohepatitis (NASH) patients: a connection between endogenous alcohol and NASH. Hepatology. 2013 Feb;57(2):601-9. doi: 10.1002/hep.26093. Epub 2013 Jan 8. PMID 23055155
- [Background] Wong VW, Tse CH, Lam TT, Wong GL, Chim AM, Chu WC, Yeung DK, Law PT, Kwan HS, Yu J, Sung JJ, Chan HL. Molecular characterization of the fecal microbiota in patients with nonalcoholic steatohepatitis--a longitudinal study. PLoS One. 2013 Apr 25;8(4):e62885. doi: 10.1371/journal.pone.0062885. Print 2013. PMID 23638162
- [Background] Karlsson FH, Fak F, Nookaew I, Tremaroli V, Fagerberg B, Petranovic D, Backhed F, Nielsen J. Symptomatic atherosclerosis is associated with an altered gut metagenome. Nat Commun. 2012;3:1245. doi: 10.1038/ncomms2266. PMID 23212374
- [Background] Glicksman C, Pournaras DJ, Wright M, Roberts R, Mahon D, Welbourn R, Sherwood R, Alaghband-Zadeh J, le Roux CW. Postprandial plasma bile acid responses in normal weight and obese subjects. Ann Clin Biochem. 2010 Sep;47(Pt 5):482-4. doi: 10.1258/acb.2010.010040. Epub 2010 Jul 1. PMID 20595403
- [Background] Vincent RP, Omar S, Ghozlan S, Taylor DR, Cross G, Sherwood RA, Fandriks L, Olbers T, Werling M, Alaghband-Zadeh J, le Roux CW. Higher circulating bile acid concentrations in obese patients with type 2 diabetes. Ann Clin Biochem. 2013 Jul;50(Pt 4):360-4. doi: 10.1177/0004563212473450. Epub 2013 Jun 14. PMID 23771134
- [Background] Watanabe M, Horai Y, Houten SM, Morimoto K, Sugizaki T, Arita E, Mataki C, Sato H, Tanigawara Y, Schoonjans K, Itoh H, Auwerx J. Lowering bile acid pool size with a synthetic farnesoid X receptor (FXR) agonist induces obesity and diabetes through reduced energy expenditure. J Biol Chem. 2011 Jul 29;286(30):26913-20. doi: 10.1074/jbc.M111.248203. Epub 2011 Jun 1. PMID 21632533
- [Background] Ma Y, Huang Y, Yan L, Gao M, Liu D. Synthetic FXR agonist GW4064 prevents diet-induced hepatic steatosis and insulin resistance. Pharm Res. 2013 May;30(5):1447-57. doi: 10.1007/s11095-013-0986-7. Epub 2013 Feb 1. PMID 23371517
- [Background] Teodoro JS, Rolo AP, Palmeira CM. Hepatic FXR: key regulator of whole-body energy metabolism. Trends Endocrinol Metab. 2011 Nov;22(11):458-66. doi: 10.1016/j.tem.2011.07.002. Epub 2011 Aug 19. PMID 21862343
- [Background] Mudaliar S, Henry RR, Sanyal AJ, Morrow L, Marschall HU, Kipnes M, Adorini L, Sciacca CI, Clopton P, Castelloe E, Dillon P, Pruzanski M, Shapiro D. Efficacy and safety of the farnesoid X receptor agonist obeticholic acid in patients with type 2 diabetes and nonalcoholic fatty liver disease. Gastroenterology. 2013 Sep;145(3):574-82.e1. doi: 10.1053/j.gastro.2013.05.042. Epub 2013 May 30. PMID 23727264
- [Background] Keitel V, Haussinger D. Perspective: TGR5 (Gpbar-1) in liver physiology and disease. Clin Res Hepatol Gastroenterol. 2012 Oct;36(5):412-9. doi: 10.1016/j.clinre.2012.03.008. Epub 2012 Apr 18. PMID 22521118
- [Background] Svensson PA, Olsson M, Andersson-Assarsson JC, Taube M, Pereira MJ, Froguel P, Jacobson P. The TGR5 gene is expressed in human subcutaneous adipose tissue and is associated with obesity, weight loss and resting metabolic rate. Biochem Biophys Res Commun. 2013 Apr 19;433(4):563-6. doi: 10.1016/j.bbrc.2013.03.031. Epub 2013 Mar 22. PMID 23523790
- [Background] Shalhub S, Parsee A, Gallagher SF, Haines KL, Willkomm C, Brantley SG, Pinkas H, Saff-Koche L, Murr MM. The importance of routine liver biopsy in diagnosing nonalcoholic steatohepatitis in bariatric patients. Obes Surg. 2004 Jan;14(1):54-9. doi: 10.1381/096089204772787293. PMID 14980034
- [Background] Lima ML, Mourao SC, Diniz MT, Leite VH. Hepatic histopathology of patients with morbid obesity submitted to gastric bypass. Obes Surg. 2005 May;15(5):661-9. doi: 10.1381/0960892053923888. PMID 15946458
- [Background] Helling TS, Helzberg JH, Nachnani JS, Gurram K. Predictors of nonalcoholic steatohepatitis in patients undergoing bariatric surgery: when is liver biopsy indicated? Surg Obes Relat Dis. 2008 Sep-Oct;4(5):612-7. doi: 10.1016/j.soard.2007.11.007. Epub 2008 Jan 28. PMID 18226970
- [Background] Dolce CJ, Russo M, Keller JE, Buckingham J, Norton HJ, Heniford BT, Gersin KS, Kuwada TS. Does liver appearance predict histopathologic findings: prospective analysis of routine liver biopsies during bariatric surgery. Surg Obes Relat Dis. 2009 May-Jun;5(3):323-8. doi: 10.1016/j.soard.2008.12.008. Epub 2009 Jan 23. PMID 19356994
- [Background] Teixeira AR, Bellodi-Privato M, Carvalheira JB, Pilla VF, Pareja JC, D'Albuquerque LA. The incapacity of the surgeon to identify NASH in bariatric surgery makes biopsy mandatory. Obes Surg. 2009 Dec;19(12):1678-84. doi: 10.1007/s11695-009-9980-x. PMID 19789933
- [Background] Junior WS, Nonino-Borges CB. Clinical predictors of different grades of nonalcoholic fatty liver disease. Obes Surg. 2012 Feb;22(2):248-52. doi: 10.1007/s11695-011-0438-6. PMID 21598007
- [Background] Ramos-De la Medina A, Remes-Troche JM, Roesch-Dietlen FB, Perez-Morales AG, Martinez S, Cid-Juarez S. Routine liver biopsy to screen for nonalcoholic fatty liver disease (NAFLD) during cholecystectomy for gallstone disease: is it justified? J Gastrointest Surg. 2008 Dec;12(12):2097-102; discussion 2102. doi: 10.1007/s11605-008-0704-7. Epub 2008 Sep 30. PMID 18825466
- [Background] Ruhl CE, Everhart JE. Relationship of non-alcoholic fatty liver disease with cholecystectomy in the US population. Am J Gastroenterol. 2013 Jun;108(6):952-8. doi: 10.1038/ajg.2013.70. Epub 2013 Apr 2. PMID 23545713
- [Background] Nervi F, Arrese M. Cholecystectomy and NAFLD: does gallbladder removal have metabolic consequences? Am J Gastroenterol. 2013 Jun;108(6):959-61. doi: 10.1038/ajg.2013.84. PMID 23735917
- [Background] Amigo L, Husche C, Zanlungo S, Lutjohann D, Arrese M, Miquel JF, Rigotti A, Nervi F. Cholecystectomy increases hepatic triglyceride content and very-low-density lipoproteins production in mice. Liver Int. 2011 Jan;31(1):52-64. doi: 10.1111/j.1478-3231.2010.02361.x. Epub 2010 Oct 29. PMID 21040411
- [Background] Mande SS, Mohammed MH, Ghosh TS. Classification of metagenomic sequences: methods and challenges. Brief Bioinform. 2012 Nov;13(6):669-81. doi: 10.1093/bib/bbs054. Epub 2012 Sep 8. PMID 22962338